CLINICAL TRIAL: NCT06250868
Title: TRK-3 Agreement and Precision of Pachymetry Function
Brief Title: TRK-3 Performance of Pachymetry
Status: Completed | Type: Observational
Sponsor: Topcon Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: THQ-THINC-2023-03
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Normal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Normal cornea
  Interventions: Device: Kerato-Refracto Tonometer

INTERVENTIONS:
Device: Kerato-Refracto Tonometer — measures pressure inside the eye and thickness of the cornea.

SUMMARY:
To evaluate the performance of a new tonometer.

ELIGIBILITY:
Inclusion Criteria:

1. Provide voluntary written consent for participation in the study.
2. Age at least 22 years old at the time of informed consent.

Exclusion Criteria:

1. Ocular condition that may affect the ability to perform corneal measurement (e.g., corneal perforation, bullous keratopathy, nystagmus)
2. Have or is suspected to have an ocular infection in either eye.
3. Otherwise considered unsuitable for the study by the investigator
4. Unable to tolerate ophthalmic testing.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who have healthy cornea
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
Cornea thickness | 1 day
  Thickness of the cornea

CONTACTS AND LOCATIONS:
Locations (1):
- Topcon Healthcare Innovation Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No